CLINICAL TRIAL: NCT02958774
Title: Hypofractionated Radiation Therapy for Patients With Breast Cancer Receiving Regional Nodal Irradiation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-MM-BRST-HypoFracRT
Record Dates: First submitted 2016-09-30; First posted 2016-11-08 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypofractionated Radiation Therapy (Experimental): Daily for 4 weeks
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Chest/Breast 4005 centigray (cGy)/15 fractions/267 cGy daily Regional nodes 4005 cGy/15 fractions/267 cGy daily 1000 cGy boost to lumpectomy/scar/undissected nodes 200 cGy daily

SUMMARY:
The primary objective of this study is to document lymphedema rates in patients requiring regional nodal irradiation (RNI) who receive hypofractionated radiation as compared to conventional radiation.

DETAILED DESCRIPTION:
Participants with stage II or stage III node-positive breast cancer, or T3N0 node-negative will receive hypofractionated radiation for 4 weeks. We hypothesize that patients receiving a shorter course of radiation will have reduced lymphedema. Lymphedema is diagnosed when the patient's arm circumference measures 10% or more as compared to pre-treatment (baseline) arm circumference measurement. Secondary endpoints will address the effectiveness, quality of life, and side effect profile of a shortened course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Status 50% - 100%
* Diagnosis of stage II or III node-positive breast cancer (NOTE: Stages include: T4a-cNany, T3N1, TxN2.) OR T3N0 node-negative breast cancer.
* For patients with TxN1 disease, one of the following criteria must be met: Grade 3; ≤ 45 years of age at time of screening for this study; extensive Lymphovascular Space Invasion (LVSI); 3 lymph nodes positive; hormone-negative disease; positive lymph nodes after chemotherapy; or extracapsular extension
* Prior surgery and chemotherapy allowed, no prior radiation to the target area (breast or chest and nodes). NOTE: Radiation should occur 3-12 weeks after last chemotherapy or surgery, whichever comes last.
* Women of child-bearing potential (WOCP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

Exclusion Criteria:

* Diagnosis of inflammatory breast cancer
* Previously diagnosed malignancy excluding basal or squamous cell carcinoma of the skin (unless disease-free for 5 years or more)
* Diagnosis of scleroderma
* Diagnosis of lupus
* Diagnosis of active dermatomyositis
* Diagnosis of metastatic disease
* Pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Lymphedema Rate | One year post end of treatment (EOT)
  Defined as a 10% increase in arm circumference from pre-treatment (baseline) arm circumference measurement.

SECONDARY OUTCOMES:
Local Recurrence | 12 months post-EOT
  Defined as biopsy proven recurrence of breast cancer involving the chest wall, breast, axilla, internal mammary or supraclavicular nodes
Cosmetic (Breast) Outcome | 12 months post-EOT
  Measured using the Breast Q™ Assessment questionnaire
Quality of Life | After enrollment but prior to CT simulation; 14-90 days post-EOT; 12 months post-EOT
  Measured using the Functional Assessment of Cancer Therapy Questionnaire for Breast Cancer (FACT-B+4) questionnaire
Range of Motion (Upper Extremities) | 14-90 days post-EOT; 6 months post-EOT; 12 months post-EOT
  Percent reduction in referrals to physical therapy for impaired range of movement post-EOT

CONTACTS AND LOCATIONS:
Overall Officials: Shane Stecklein, MD, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States